CLINICAL TRIAL: NCT01923753
Title: A Short-term Comparative Study of Aerosure for Airway Clearance in Patients With Cystic Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit sufficient patients within reasonable timeframe
Sponsor: Actegy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ACACIA-01
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Neural respiratory drive; Airway clearance technique; Expectoration; Positive expiratory pressure device
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aerosure 15 Hz (Experimental): All subjects receive an active device operating at a specific frequency, active device operating at another specific frequency and sham device (disabled):
  Aerosure at 15 Hz; Aerosure at 25 Hz; Sham Aerosure. Order of presentation is randomised.
  Interventions: Device: Aerosure at 15 Hz
- Aerosure 25 Hz (Active Comparator): All subjects receive an active device operating at a specific frequency, active device operating at another specific frequency and sham device (disabled):
  Aerosure at 15 Hz; Aerosure at 25 Hz; Sham Aerosure.
  Interventions: Device: Aerosure at 25 Hz
- Aerosure sham (Sham Comparator): All subjects receive an active device operating at a specific frequency, active device operating at another specific frequency and sham device (disabled):
  Aerosure at 15 Hz; Aerosure at 25 Hz; Sham Aerosure.
  Interventions: Device: Sham Aerosure

INTERVENTIONS:
Device: Aerosure at 15 Hz — Active Aerosure HFAO device operating at lower frequency
  Arms: Aerosure 15 Hz
Device: Aerosure at 25 Hz — Active Aerosure HFAO device operating at higher frequency
  Arms: Aerosure 25 Hz
Device: Sham Aerosure — Deactivated but identical Aerosure HFAO device
  Arms: Aerosure sham

SUMMARY:
This is a double-blind randomised controlled crossover study to investigate whether high frequency airflow oscillation (HFAO), delivered using Aerosure, improves sputum clearance in patients admitted to hospital with infective exacerbations of cystic fibrosis (CF). This study will test the hypothesis that the wet weight of sputum expectorated is greater following the use of Aerosure than following the use of a sham Aerosure device.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CF (established by genotype or sweat sodium >70mmol/l or sweat chloride of >60 mmol/l
* Admitted to King's College Hospital within 48 hours of an acute infective pulmonary exacerbation characterised by an increase in respiratory symptoms requiring intravenous antibiotics

Exclusion Criteria:

* Acute respiratory failure
* Haemodynamic instability (including severe right heart failure with hypotension)
* Current severe haemoptysis
* Ineffective cough
* Rib fractures
* Pregnancy
* Current or recent pneumothorax
* Epilepsy
* Current pulmonary embolism
* Oesophageal varices
* Recent thoracic upper gastro-intestinal tract or facial surgery
* Active tuberculosis
* Recent brain, eye, ear, ENT surgery
* Myocardial infarction
* Ascending aortic aneurysm
* Acute diarrhoea
* Pulmonary embolism
* Angina
* Severe hypertension (systolic >200 mm Hg, diastolic >120 mm Hg)
* Confusion/dementia
* Inability to give consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Wet weight of sputum expectorated during treatment session | up to 30 minutes after treatment

SECONDARY OUTCOMES:
Change in FEV1 | immediately before and up to 30 minutes after treatment
Change in VC | immediately before and up to 30 minutes after treatment
Change in oxygen saturation | continuously from 3 minutes prior to treatment and until 3 minutes after treatment
Change in ventilation | 5 minutes prior to treatment, immediately following treatment and 30 minutes after treatment
Change in neural respiratory drive | 5 minutes prior to treatment and 30 minutes after treatment

CONTACTS AND LOCATIONS:
Overall Officials: John Moxham, MD, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital, Bessemer Road, Denmark Hill, London, United Kingdom